CLINICAL TRIAL: NCT01130831
Title: A Phase IV, Multi-Centre, Non-interventional Study Evaluating the Effect of Lanthanum Carbonate in Patients Previously Treated With Calcium Based Phosphate Binder Therapy on Serum Phosphorous Control, Concomitant Vitamin D Therapy and Bone Related Biochemical Parameters in End Stage Renal Disease Patients on Hemodialysis
Brief Title: Effect of Lanthanum Carbonate in Patients Previously Treated With Calcium-based Phosphate Binder Therapy
Status: Completed | Type: Observational
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Other Study IDs: SPD405-702
Record Dates: First submitted 2010-05-20; First posted 2010-05-26 (Estimated); Results first posted 2013-07-04 (Estimated); Last update posted 2021-06-28 (Actual); Status verified 2021-06

CONDITIONS: End Stage Renal Disease
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — lanthanum carbonate

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

INTERVENTIONS:
Drug: Lanthanum carbonate
  Other Names: Fosrenol

SUMMARY:
To assess the percentage of patients on lanthanum carbonate, that achieve Kidney Disease Outcome Quality Initiative (KDOQI) guideline suggested values for serum phosphorous in patients previously treated with calcium-based phosphate binder therapy.

ELIGIBILITY:
Inclusion Criteria:

Patients meeting all of the criteria listed below may be included in the study:

1. Patients aged over 18 years
2. Patients with ESRD on haemodialysis who are willing and able to provide written informed consent.
3. Patients on:

   * Lanthanum carbonate monotherapy for ≥1 month
   * Lanthanum carbonate monotherapy for ≤3 months
   * Calcium-based monotherapy for ≥3 months immediately prior to lanthanum carbonate therapy.
4. Values recorded in medical records detailing serum phosphorous, serum calcium-phosphorus product, iPTH, and medication ≤6 months prior to commencing lanthanum carbonate therapy and whilst on a calcium-based monotherapy.

Exclusion Criteria:

Patients are excluded from the study if any of the following criteria are met at screening:

1. Known or suspected intolerance or hypersensitivity to lanthanum, or any of the stated ingredients
2. Patients with known hypophosphatemia (phosphate level below lower level of normal)
3. Patients with severe hepatic impairment
4. Patients with requirement for calcium supplementation for reasons other than CKD
5. Pregnant or lactating women and women planning to become pregnant over the next 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Haemodialysis patients with hyperphosphataemia
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2010-04-26 (Actual); Primary Completion 2012-06-12 (Actual); Study Completion 2012-06-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (31):
- Germany (31):
  - Dialysezentrum Facharzt für Innere Medizin und Nephrologie, Homberg (Ohm), Hesse
  - Dialyse Alsfeld, Alsfeld
  - Nephrologische Praxis Altötting-Burghausen, Altötting
  - Dialyse am Treptower Park, Berlin
  - Dialyse Berlin, Berlin
  - Dialysezentrum Cochem, Cochem
  - Dialysezentrum Coesfeld, Coesfeld
  - MVZ Caspar-David-Friedrich-Str., Dresden
  - Dialysezentrum Karlstraße, Düsseldorf
  - Dialysezentrum Süd, Düsseldorf
  - KfH-Nierenzentrum Eberswalde, Eberswalde
  - Arzt für Dialyse, Facharzt für Innere Medizin und Nephrologie, Essen
  - Dialysezentrum Lauerwald, Gera
  - Dialysezentrum Grevenbroich, Grevenbroich
  - Dialyse im Heidering, Hanover
  - Dialysepraxen Herne und Wanne-Eickel, Herne
  - Dialyse Herzberg, Herzberg
  - Patienten-Heimversorgung, Hildesheim
  - Universitätsklinik des Saarlandes, Homburg / Saar
  - Nierenzentrum Mannheim, Mannheim
  - Dialysepraxis, Meiningen
  - Dialyse Mettmann, Mettmann
  - Nierenzentrum Bogenhausen, München
  - Nephrologie Nettetal, Nettetal
  - Dialysenzentrum Peine, Peine
  - Facharzt für Innere Medizin und Nephrologie, Potsdam
  - Facharzt für Innere Medizin und Nephrologie, Quedlinburg
  - Nephrologische Praxis Schwetzingen, Schwetzingen
  - PHV-Dialysezentrum Siegen, Siegen
  - Nephrologisches Zentrum, Villingen-Schwenningen
  - Dialysezentrum Worms, Worms

RESULTS

PARTICIPANT FLOW:
Groups:
- Lanthanum Carbonate: Lanthanum carbonate therapy after previous calcium-based phosphate binder therapy treatment for >=3 months.
Period: Overall Study
Arm/Group | Lanthanum Carbonate
Started | 66
Completed | 52
Not Completed | 14
Not completed — Withdrawal by Subject | 7
Not completed — Death | 4
Not completed — Information was missing | 3

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set included all screened subjects who took at least 1 dose of lanthanum carbonate and for whom 1 follow-up assessment was completed (n = 61).
Arm/Group | Lanthanum Carbonate
Number analyzed (Participants) | 61
Age, Continuous [Mean (Standard Deviation); unit: years] — Safety Analysis Set
  years | 66.0 (12.5)
Age, Customized [Count of Participants; unit: Participants] — Safety Analysis Set
  Participants
    >=18 years | 61
Sex: Female, Male [Count of Participants; unit: Participants] — Safety Analysis Set
  Participants
    Female | 22
    Male | 39
Region of Enrollment [Count of Participants; unit: Participants] — Safety Analysis Set
  Participants
    Germany | 61

OUTCOME MEASURES:

1. Primary Outcome: Percent of Subjects That Achieved Controlled Serum Phosphorous Levels on Calcium-based Phosphate Binder Therapy
Description: Phosphorous levels are controlled if they meet the Kidney Disease Outcomes Quality Initiative (KDOQI) target for serum phosphorous of 3.5-5.5 mg/dL.
Time Frame: Baseline
Population: Full Analysis Set included subjects of the Safety Analysis Set who had values for serum phosphorous, serum calcium, and intact parathyroid hormone (iPTH) while on prior calcium-based phosphate binder therapy.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Groups:
- Calcium-based Phosphate Binder Therapy: The percent of subjects that achieved the serum phosphate KDOQI target on previous calcium-based phosphate binder therapy of >=3 months of treatment prior to receiving lanthanum carbonate treatment.
Arm/Group | Calcium-based Phosphate Binder Therapy
Number analyzed (Participants) | 47
percentage of subjects | 14.9 [6.2 to 28.3]

2. Secondary Outcome: Percent of Subjects That Achieved Controlled Serum Calcium Levels on Calcium-based Phosphate Binder Therapy
Description: Calcium levels are controlled if they meet the Kidney Disease Outcomes Quality Initiative (KDOQI) target for serum calcium of 8.4-9.5 mg/dL.
Time Frame: Baseline
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Groups:
- Calcium-based Phosphate Binder Therapy: The percent of subjects that achieved the serum calcium KDOQI target on previous calcium-based phosphate binder therapy for >=3 months prior to receiving lanthanum carbonate treatment.
Arm/Group | Calcium-based Phosphate Binder Therapy
Number analyzed (Participants) | 47
percentage of subjects | 68.1 [52.9 to 80.9]

3. Secondary Outcome: Percent of Subjects That Achieved Controlled Serum Calcium Levels on Lanthanum Carbonate Therapy
Description: as for outcome 2
Time Frame: 12 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Groups:
- Lanthanum Carbonate: The percent of subjects that achieved the serum calcium KDOQI target on lanthanum carbonate after previous calcium-based phosphate binder therapy treatment for >=3 months.
Arm/Group | Lanthanum Carbonate
Number analyzed (Participants) | 40
percentage of subjects | 52.5 [36.1 to 68.5]

4. Secondary Outcome: Percent of Subjects That Achieved Controlled Serum Calcium-Phosphorous Product Levels on Calcium-based Phosphate Binder Therapy
Description: Calcium-phosphorous product levels are controlled if they meet the Kidney Disease Outcomes Quality Initiative (KDOQI) target for serum calcium-phosphorous product of <55 mg^2/dL^2.
Time Frame: Baseline
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Groups:
- Calcium-based Phosphate Binder Therapy: The percent of subjects that achieved the serum calcium-phosphorous product KDOQI target on previous calcium-based phosphate binder therapy for >=3 months prior to receiving lanthanum carbonate treatment.
Arm/Group | Calcium-based Phosphate Binder Therapy
Number analyzed (Participants) | 47
percentage of subjects | 42.6 [28.3 to 57.8]

5. Secondary Outcome: Percent of Subjects That Achieved Controlled Serum Calcium-Phosphorous Product Levels on Lanthanum Carbonate Therapy
Description: as for outcome 4
Time Frame: 12 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Groups:
- Lanthanum Carbonate: The percent of subjects that achieved the serum calcium-phosphorous product levels KDOQI target on lanthanum carbonate after previous calcium-based phosphate binder therapy treatment for >=3 months.
Arm/Group | Lanthanum Carbonate
Number analyzed (Participants) | 40
percentage of subjects | 75.0 [58.8 to 87.3]

6. Secondary Outcome: Percent of Subjects That Maintained Control of Serum Phosphorous Levels on Lanthanum Carbonate
Description: as for outcome 1
Time Frame: 12 months
Population: as for outcome 1
Measure: Number; unit: percentage of subjects
Groups:
- Lanthanum Carbonate: The percent of subjects that maintained the serum phosphorous KDOQI target on lanthanum carbonate.
Arm/Group | Lanthanum Carbonate
Number analyzed (Participants) | 42
percentage of subjects
  <=1 quarter | 73.8
  2 consecutive quarters | 7.1
  3 consecutive quarters | 7.1
  4 consecutive quarters | 11.9

7. Secondary Outcome: Percent of Subjects That Maintained Control of Serum Calcium Levels on Lanthanum Carbonate
Description: as for outcome 2
Time Frame: 12 months
Population: as for outcome 1
Measure: Number; unit: percentage of subjects
Groups:
- Lanthanum Carbonate: The percent of subjects that maintained the serum calcium KDOQI target on lanthanum carbonate.
Arm/Group | Lanthanum Carbonate
Number analyzed (Participants) | 41
percentage of subjects
  <=1 quarter | 53.7
  2 consecutive quarters | 22.0
  3 consecutive quarters | 7.3
  4 consecutive quarters | 17.1

8. Secondary Outcome: Percent of Subjects That Maintained Control of Serum Calcium-Phosphorous Product Levels on Lanthanum Carbonate Therapy
Description: as for outcome 4
Time Frame: 12 months
Population: as for outcome 1
Measure: Number; unit: percentage of subjects
Groups:
- Lanthanum Carbonate: The percent of subjects that maintained the serum calcium-phosphorous product KDOQI target on lanthanum carbonate.
Arm/Group | Lanthanum Carbonate
Number analyzed (Participants) | 40
percentage of subjects
  <=1 quarter | 47.5
  2 consecutive quarters | 17.5
  3 consecutive quarters | 5.0
  4 consecutive quarters | 30.0

9. Primary Outcome: Percent of Subjects That Achieved Controlled Serum Phosphorous Levels on Lanthanum Carbonate
Description: as for outcome 1
Time Frame: 12 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Groups:
- Lanthanum Carbonate: The percent of subjects that achieved the serum phosphate KDOQI target on lanthanum carbonate after previous calcium-based phosphate binder therapy treatment for >=3 months.
Arm/Group | Lanthanum Carbonate
Number analyzed (Participants) | 40
percentage of subjects | 40.0 [24.9 to 56.7]

10. Secondary Outcome: Percent of Subjects That Maintained Control of Intact Parathyroid Hormone (iPTH) Levels on Lanthanum Carbonate Therapy
Description: iPTH levels are controlled if they meet the Kidney Disease Outcomes Quality Initiative (KDOQI) target for iPTH of 150-300 pg/mL
Time Frame: 12 months
Population: as for outcome 1
Measure: Number; unit: percentage of subjects
Groups:
- Lanthanum Carbonate: The percent of subjects that maintained the iPTH KDOQI target on lanthanum carbonate.
Arm/Group | Lanthanum Carbonate
Number analyzed (Participants) | 38
percentage of subjects
  <=1 quarter | 81.6
  2 consecutive quarters | 10.5
  3 consecutive quarters | 2.6
  4 consecutive quarters | 5.3

11. Secondary Outcome: Percent Change From Baseline in Phosphorous Levels at 12 Months
Time Frame: Baseline and 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent change in phosphorous levels
Arm/Group | Lanthanum Carbonate
Number analyzed (Participants) | 40
percent change in phosphorous levels | -7.9 (24.3)

12. Secondary Outcome: Percent Change From Baseline in Calcium Levels at 12 Months
Time Frame: Baseline and 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent change in calcium levels
Arm/Group | Lanthanum Carbonate
Number analyzed (Participants) | 40
percent change in calcium levels | -1.1 (8.1)

13. Secondary Outcome: Percent Change From Baseline in Calcium-Phosphorous Product Levels at 12 Months
Time Frame: Baseline and 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent change in calcium-phosphorous
Arm/Group | Lanthanum Carbonate
Number analyzed (Participants) | 40
percent change in calcium-phosphorous | -8.7 (26.5)

14. Secondary Outcome: Percent Change From Baseline in iPTH Levels at 12 Months
Time Frame: Baseline and 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent change in iPTH levels
Arm/Group | Lanthanum Carbonate
Number analyzed (Participants) | 32
percent change in iPTH levels | 95.4 (393.4)

15. Secondary Outcome: Percent Change From Baseline in 25-Hydroxy Vitamin D Levels at 12 Months
Time Frame: Baseline and 12 months
Population: Full Analysis Set included subjects of the Safety Analysis Set who had values for serum phosphorous, serum calcium, and intact parathyroid hormone (iPTH) while on prior calcium-based phosphate binder therapy. Note that there are a high number of missing values (n=36) for this outcome which does not allow for any meaningful comparison.
Measure: Mean (Standard Deviation); unit: percent change in vitamin D
Arm/Group | Lanthanum Carbonate
Number analyzed (Participants) | 6
percent change in vitamin D | 41.0 (48.6)

16. Secondary Outcome: Percent Change From Baseline in 1,25-Hydroxy Vitamin D Levels at 12 Months
Time Frame: Baseline and 12 months
Population: Full Analysis Set included subjects of the Safety Analysis Set who had values for serum phosphorous, serum calcium, and intact parathyroid hormone (iPTH) while on prior calcium-based phosphate binder therapy. Note that there are a high number of missing values (n=38) for this outcome which does not allow for any meaningful comparison.
Measure: Mean (Standard Deviation); unit: percent change in vitamin D
Arm/Group | Lanthanum Carbonate
Number analyzed (Participants) | 4
percent change in vitamin D | 1.1 (28.6)

17. Secondary Outcome: Percent of Subjects With Hypocalcemic Events on Calcium-based Phosphate Binder Therapy
Description: Hypocalcemia is defined as serum calcium levels below 8.02 mg/dL
Time Frame: Baseline
Population: as for outcome 1
Measure: Number; unit: percentage of subjects
Groups:
- Calcium-based Phosphate Binder Therapy: Calcium-based phosphate binder therapy of >=3 months of treatment.
Arm/Group | Calcium-based Phosphate Binder Therapy
Number analyzed (Participants) | 47
percentage of subjects | 10.6

18. Secondary Outcome: Percent of Subjects With Hypocalcemic Events on Lanthanum Carbonate
Description: Hypocalcemia is defined as serum calcium levels below 8.02 mg/dL
Time Frame: 12 months
Population: as for outcome 1
Measure: Number; unit: percentage of subjects
Arm/Group | Lanthanum Carbonate
Number analyzed (Participants) | 40
percentage of subjects | 22.5

19. Secondary Outcome: Percent of Subjects With Hypercalcemic Events on Calcium-based Phosphate Binder Therapy
Description: Hypercalcemia is defined as total serum calcium level above 11.22 mg/dL.
Time Frame: Baseline
Population: as for outcome 1
Measure: Number; unit: percentage of subjects
Groups:
- Calcium-based Phosphate Binder Therapy: Calcium-based phosphate binder therapy for >=3 months prior.
Arm/Group | Calcium-based Phosphate Binder Therapy
Number analyzed (Participants) | 47
percentage of subjects | 0.0

20. Secondary Outcome: Percent of Subjects With Hypercalcemic Events on Lanthanum Carbonate
Description: Hypercalcemia defined as total serum calcium above 11.22 mg/dL
Time Frame: 12 months
Population: as for outcome 1
Measure: Number; unit: percentage of subjects
Arm/Group | Lanthanum Carbonate
Number analyzed (Participants) | 40
percentage of subjects | 0.0

21. Secondary Outcome: Change From Baseline in Vitamin D Dose at 12 Months
Time Frame: Baseline and 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng
Arm/Group | Lanthanum Carbonate
Number analyzed (Participants) | 33
ng | -0.7 (0.0075)

22. Secondary Outcome: Change From Baseline in Mean Total Daily Dose of Calcium at 12 Months
Time Frame: Baseline and 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Lanthanum Carbonate
Number analyzed (Participants) | 6
mg | -178.6 (437.6)

23. Secondary Outcome: Number of Tablets Per Day
Time Frame: 12 months
Population: Full Analysis Set included subjects of the Safety Analysis Set who had values for serum phosphorous, serum calcium, and intact parathyroid hormone (iPTH) while on prior
Measure: Mean (Standard Deviation); unit: Number of Tablets
Arm/Group | Lanthanum Carbonate
Number analyzed (Participants) | 35
Number of Tablets | 3.4 (1.3)

ADVERSE EVENTS:
Description: Safety Analysis Set (n = 61)
Arm/Group | Lanthanum Carbonate
Serious Adverse Events (participants affected / at risk) | 0/61
Other Adverse Events (participants affected / at risk) | 0/61

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.